CLINICAL TRIAL: NCT00129974
Title: A Phase II Trial of Pemetrexed in Combination With Gemcitabine as First Line Treatment in Extensive-Stage Small Cell Lung Carcinoma
Brief Title: Study of Pemetrexed and Gemcitabine for Patients With a New Diagnosis of Extensive-Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: failure to accrue
Sponsor: Tufts Medical Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7338
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Small Cell
Keywords: Lung cancer; Phase II; Drug Therapy
MeSH Terms: conditions — Carcinoma, Small Cell; Lung Neoplasms | interventions — Pemetrexed; Gemcitabine

INTERVENTIONS:
Drug: pemetrexed and gemcitabine

SUMMARY:
The purpose of the study is to determine whether pemetrexed and gemcitabine cause good tumour shrinkage when given to patients with previously untreated extensive-stage small cell lung cancer. The second purpose is to see if the side effects appear better than what is expected with standard chemotherapy.

DETAILED DESCRIPTION:
Extensive-stage small cell lung carcinoma is incurable. Present therapies are toxic and responses are short lived. This phase II, single arm, window of opportunity study will assess the response rate and toxicity of pemetrexed and gemcitabine in this cohort.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of extensive small cell lung cancer. For this study, extensive stage disease will be defined as including those patients whose disease cannot be encompassed in a curative radiation field. While this definition varies by treating center, it will include patients with metastatic disease to contralateral lung parenchyma or other organs (e.g. liver) and may include patients with contralateral supraclavicular, mediastinal, or hilar lymph nodes or a pleural effusion.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral computed tomography (CT) scan.
* No history of prior chemotherapy or experimental therapy for extensive or recurrent small cell lung cancer (SCLC). Subjects may have received chemotherapy as part of treatment for limited disease, but such chemotherapy must have been completed at least 6 months prior to the diagnosis of recurrent disease.
* Prior radiation therapy is permitted if acute side effects have resolved; if the site of radiation was not the only measurable tumor site; and if less than 25% of the bone marrow was treated.
* Age > 18 years. Because no dosing or adverse event data are currently available on the use of pemetrexed in combination with gemcitabine in patients <18 years of age, children are excluded from this study.
* ECOG performance status 0-1.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes > 3,000/uL;
  * absolute neutrophil count > 1,500/uL;
  * platelets > 100,000/uL;
  * total bilirubin < 1.5 X institutional limits;
  * AST (SGOT)/ALT (SGPT) < 2 X institutional limits OR < 3 times the upper limit of normal in the presence of liver metastases;
  * serum sodium > 125 mEq/L and no syndrome of inappropriate antidiuretic hormone secretion (SIADH);
  * creatinine within normal institutional limits; AND
  * creatinine clearance > 45 mL/min by the Cockroft and Gault formula for patients with creatinine levels above institutional normal.
* Brain metastases are permitted if radiation has been administered, the subject has recovered, and corticosteroids are not required.
* The effects of pemetrexed and gemcitabine on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because anti-folate agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pemetrexed or gemcitabine.
* Pleural effusion, unless it is small, is asymptomatic, or a thoracentesis can be performed to render it small and asymptomatic prior to enrollment. Patients with significant ascites are ineligible.
* Evidence of superior vena cava syndrome or the threat of imminent obstruction of central vessels or major airways.
* Extensive liver involvement with tumor such that any significant degree of progression would increase the subject's risk of morbidity or mortality.
* A major, symptomatic, paraneoplastic syndrome such as SIADH, Eaton-Lambert, Cushing's syndrome, encephalomyelitis, etc.
* A history of prior or concurrent malignancy other than in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or other malignancy treated > 5 years previously without evidence of recurrence.
* Significant comorbidity that in the judgement of the investigator would increase the subject's risk of toxicity or death while on study.
* Pregnant women are excluded from this study because pemetrexed is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pemetrexed or gemcitabine, breastfeeding should be discontinued if the mother is treated with either agent.
* Candidates who are unwilling or unable to take vitamin supplementation or dexamethasone as outlined in the protocol; or who are unwilling or unable to interrupt nonsteroidal anti-inflammatories and salicylates (ASA) as outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-08; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Goffin, MD FRCPC, Principal Investigator — Tufts Medical Center; John McCann, MD, Principal Investigator — Baystate Medical Center; Walter A Kagan, MD PhD, Principal Investigator — Commonwealth Hematology/Oncology
Locations (3):
- United States (3):
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Commonwealth Hematology/Oncology, Quincy, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts

REFERENCES:
- See also: Baystate Cancer Center — http://baystatehealth.org/Baystate/Main+Nav/Clinical+Services/Departments/Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Pemetrexed and Gemcitabine
Period: Overall Study
Arm/Group | Arm 1
Started | 1
Completed | 0
Not Completed | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Study Termination
Arm/Group | Arm 1
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: Number of Participants with at least one Adverse Event
Time Frame: Study Termination
Arm/Group | Arm 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes